CLINICAL TRIAL: NCT03077737
Title: Reducing Tobacco Use Disparities Among Adults In Safety Net Community Health Centers
Brief Title: Reducing Tobacco Use Disparities Among Low-Income Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of Illinois at Chicago (Other); Northeastern Illinois University (Other)
Responsible Party: Principal Investigator, Brian Hitsman, Associate Professor of Preventive Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5U54CA203000 (NIH)
Record Dates: First submitted 2017-03-01; First posted 2017-03-13 (Actual); Results first posted 2022-01-12 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Cigarette Smoking; Nicotine Dependence
Keywords: Treatment access; Treatment utilization; Smoking cessation; Low income; Electronic health record system; Electronic referral
MeSH Terms: conditions — Cigarette Smoking; Tobacco Use Disorder; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Population health management (Experimental): Population health management for smoking cessation in low-income smokers: the Choose to Change intervention
  Interventions: Behavioral: Choose to Change
- Enhanced usual care (Active Comparator): Usual clinic-based care enhanced by an EHR system that can deliver an electronic referral for quitline treatment
  Interventions: Behavioral: Enhanced usual care

INTERVENTIONS:
Behavioral: Choose to Change — Population-based letter outreach automated via the electronic health record system and text messaging targeted to low-income smokers. Paired with automated electronic referral for proactive quitline treatment (behavioral counseling plus nicotine replacement therapy).
  Arms: Population health management
Behavioral: Enhanced usual care — Enhanced usual care based on Ask, Advise and Refer in which an electronic referral for proactive quitline treatment (behavioral counseling plus nicotine replacement therapy) is made during a clinic visit.
  Arms: Enhanced usual care

SUMMARY:
Most smokers, especially those who are poor, do not receive smoking cessation treatment during their healthcare visits. This study is evaluating a novel population health management intervention for low-income smokers. Automated via an EHR system, which is bidirectionally linked with the Illinois Tobacco Quitline, the intervention comprises a mailed letter and text messaging designed to motivate low-income patients, most of whom are not ready to quit, to accept and use proactive quitline treatment. Increased access to free effective treatment via the integration of healthcare systems and state quitline services may be especially significant in its impact on low-income smokers who are underserved and who carry a much greater burden of tobacco-related disease.

DETAILED DESCRIPTION:
An estimated 26 million smokers still receive no treatment for their smoking during their primary care visits. Given the persistent clinical system, provider, and patient barriers to addressing smoking in primary care, especially for poor populations, an electronic health record (EHR)-automated population health management approach that directly links the healthcare system with public health services to engage all smokers may increase access to effective treatment. Increased access is especially significant for low-income smokers who are underserved and who carry a disproportionate burden of tobacco-related disease. While 90% of smokers are not ready to quit, many are interested in cutting down, and smoking reduction increases the likelihood of future quit attempts and smoking cessation. Based on self-determination theory, population outreach targeted to low-income smokers that offers them the choice to either quit or cut down as a first step towards cessation may increase their engagement in and utilization of smoking cessation treatment and likelihood of achieving abstinence. This 2-group randomized controlled trial will evaluate the effectiveness of a population health management intervention for smoking cessation in low-income smokers. Participants will be 530 diverse, low-income smokers of a large Federally Qualified Health Center (FQHC) in Chicago identified using its EHR system. Automated via the EHR system, participants will be mailed a letter on behalf of their providers that encourages smoking cessation or smoking reduction as a first step to quitting (Choose to Change; N=265). The letter will be paired with 5 text messages 2-3 days apart that are designed to reinforce the central messaging of the letter ("Choose to change and make your own goal"). All components of the Choose to Change intervention will be offered in English and Spanish. Two weeks after letter mailing and automated electronic referral, participants will receive a call from the Illinois Tobacco Quitline and offered free behavioral counseling and free nicotine replacement therapy (NRT; patch, gum, or lozenge) for smoking cessation or reduction. Treatment will continue as either accepted or initiated by participants for 28 weeks. Treatment outcomes will be transmitted directly from the Quitline server to the EHR system. Choose to Change will be compared with Enhanced Usual Care (N=265), in which an electronic referral for proactive Quitline treatment is made during a clinic visit. The primary study outcomes will be treatment engagement (initial counseling call completed) at 6 weeks, utilization (one or more additional counseling calls completed) at 14 weeks, and smoking cessation (bioverified 7-day point-prevalence abstinence) at 28 weeks. An exploratory aim is to examine moderators of intervention effects. An EHR-automated population health management intervention targeted to low-income smokers could reduce critical disparities in treatment access, utilization, and cessation. If determined to be effective, the Choose to Change intervention could be readily disseminated to 11 other FQHCs in Chicago, comprising 85 clinical sites that care for almost 500,000 low-income patients.

ELIGIBILITY:
Inclusion criteria

1. Men and women who are 18 years of age or older
2. A patient who receives healthcare at one of the seven Near North Health Service Corporation community health centers in Chicago
3. Daily or weekly cigarette smoker
4. One or more healthcare visits within the past 12 months

Exclusion criteria

1. Language preference other than English or Spanish for their healthcare
2. No telephone number or address listed in the EHR system
3. Lives with another patient who is already enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Hitsman, PhD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University Feingberg School of Medicine, Dept. of Preventive Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piper ME, Baker TB, Mermelstein R, Collins LM, Fraser DL, Jorenby DE, Smith SS, Christiansen BA, Schlam TR, Cook JW, Oguss M, Fiore MC. Recruiting and engaging smokers in treatment in a primary care setting: developing a chronic care model implemented through a modified electronic health record. Transl Behav Med. 2013 Sep;3(3):253-63. doi: 10.1007/s13142-012-0178-8. PMID 24073176
- [Background] Hughes JR, Carpenter MJ. Does smoking reduction increase future cessation and decrease disease risk? A qualitative review. Nicotine Tob Res. 2006 Dec;8(6):739-49. doi: 10.1080/14622200600789726. PMID 17132521
- [Background] Williams GC, McGregor HA, Sharp D, Levesque C, Kouides RW, Ryan RM, Deci EL. Testing a self-determination theory intervention for motivating tobacco cessation: supporting autonomy and competence in a clinical trial. Health Psychol. 2006 Jan;25(1):91-101. doi: 10.1037/0278-6133.25.1.91. PMID 16448302
- [Background] Jamal A, Dube SR, Malarcher AM, Shaw L, Engstrom MC; Centers for Disease Control and Prevention (CDC). Tobacco use screening and counseling during physician office visits among adults--National Ambulatory Medical Care Survey and National Health Interview Survey, United States, 2005-2009. MMWR Suppl. 2012 Jun 15;61(2):38-45. PMID 22695462
- [Background] Boyle RG, Solberg LI, Fiore MC. Electronic medical records to increase the clinical treatment of tobacco dependence: a systematic review. Am J Prev Med. 2010 Dec;39(6 Suppl 1):S77-82. doi: 10.1016/j.amepre.2010.08.014. PMID 21074681
- [Background] Yarnall KS, Pollak KI, Ostbye T, Krause KM, Michener JL. Primary care: is there enough time for prevention? Am J Public Health. 2003 Apr;93(4):635-41. doi: 10.2105/ajph.93.4.635. PMID 12660210
- [Background] Baker DW, Parker RM, Williams MV, Clark WS, Nurss J. The relationship of patient reading ability to self-reported health and use of health services. Am J Public Health. 1997 Jun;87(6):1027-30. doi: 10.2105/ajph.87.6.1027. PMID 9224190
- [Background] Lindson-Hawley N, Aveyard P, Hughes JR. Gradual reduction vs abrupt cessation as a smoking cessation strategy in smokers who want to quit. JAMA. 2013 Jul 3;310(1):91-2. doi: 10.1001/jama.2013.6473. PMID 23821093
- [Background] Hiscock R, Bauld L, Amos A, Fidler JA, Munafo M. Socioeconomic status and smoking: a review. Ann N Y Acad Sci. 2012 Feb;1248:107-23. doi: 10.1111/j.1749-6632.2011.06202.x. Epub 2011 Nov 17. PMID 22092035
- [Background] Williams GC, Niemiec CP, Patrick H, Ryan RM, Deci EL. The importance of supporting autonomy and perceived competence in facilitating long-term tobacco abstinence. Ann Behav Med. 2009 Jun;37(3):315-24. doi: 10.1007/s12160-009-9090-y. Epub 2009 Apr 17. PMID 19373517
- [Background] Landon BE, Grumbach K, Wallace PJ. Integrating public health and primary care systems: potential strategies from an IOM report. JAMA. 2012 Aug 1;308(5):461-2. doi: 10.1001/jama.2012.8227. No abstract available. PMID 22851111
- [Derived] Hitsman B, Matthews PA, Papandonatos GD, Cameron KA, Rittner SS, Mohanty N, Long T, Ackermann RT, Ramirez E, Carr J, Cordova E, Bridges C, Flowers-Carson C, Giachello AL, Hamilton A, Ciecierski CC, Simon MA. An EHR-automated and theory-based population health management intervention for smoking cessation in diverse low-income patients of safety-net health centers: a pilot randomized controlled trial. Transl Behav Med. 2022 Oct 7;12(9):892-899. doi: 10.1093/tbm/ibac026. PMID 36205472

RESULTS

PARTICIPANT FLOW:
Period: Week 6 (10 Weeks After Enrollment)
Arm/Group | Population Health Management | Enhanced Usual Care
Started | 97 | 93
Completed | 89 | 79
Not Completed | 8 | 14
Period: Week 14 (18 Weeks After Enrollment)
Arm/Group | Population Health Management | Enhanced Usual Care
Started | 97 | 93
Completed | 83 | 76
Not Completed | 14 | 17
Period: Week 28 (32 Weeks After Enrollment)
Arm/Group | Population Health Management | Enhanced Usual Care
Started (Due to project timeline constraints, only the first 96 participants enrolled in the study were followed for 32 weeks.) | 49 | 47
Completed | 39 | 40
Not Completed | 10 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Population Health Management | Enhanced Usual Care | Total
Number analyzed (Participants) | 97 | 93 | 190
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (10.7) | 48.8 (11.9) | 49.0 (11.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Females | 58 | 65 | 123
  Males | 49 | 28 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 16
  Not Hispanic or Latino | 89 | 85 | 174
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 81 | 75 | 156
  White | 8 | 7 | 15
  More than one race | 2 | 6 | 8
  Unknown or Not Reported | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Quitline Treatment Engagement
Description: The number of participants who accepted the quitline call and accepted treatment as defined by enrolling in treatment and completing the first counseling session. Participants who returned a quitline call, enrolled in treatment, and completed the first counseling session were also counted as having engaged in treatment.
Time Frame: Week 6
Measure: Count of Participants; unit: Participants
Arm/Group | Population Health Management | Enhanced Usual Care
Number analyzed (Participants) | 97 | 93
Participants | 25 | 0

2. Primary Outcome: Quitline Treatment Utilization
Description: The number of participants who completed one or more additional quitline counseling calls.
Time Frame: Week 14
Measure: Count of Participants; unit: Participants
Arm/Group | Population Health Management | Enhanced Usual Care
Number analyzed (Participants) | 97 | 93
Participants | 21 | 0

3. Primary Outcome: Smoking Cessation at Week 28 (32 Weeks After Enrollment)
Description: Self-reported seven-day point-prevalence abstinence at week 28. Number of participants who reporting smoking cessation at week 28. Participants were classified as abstinent if they reported not smoking (not even a puff of a cigarette) for at least 7 days prior to the assessment.
Time Frame: Week 28
Population: Due to project timeline constraints, only the first 96 participants were followed for 32 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Population Health Management | Enhanced Usual Care
Number analyzed (Participants) | 49 | 47
Participants | 8 | 3

4. Secondary Outcome: Smoking Cessation at Week 14 (18 Weeks After Enrollment)
Description: Self-reported seven-day point-prevalence abstinence at week 14. Participants were classified as abstinent if they reported not smoking (not even a puff of a cigarette) for at least 7 days prior to the assessment.
Time Frame: Week 14
Measure: Count of Participants; unit: Participants
Arm/Group | Population Health Management | Enhanced Usual Care
Number analyzed (Participants) | 97 | 93
Participants | 9 | 3

ADVERSE EVENTS:
Time Frame: No adverse events were collected or assessed for this study.
Description: Not applicable. No adverse events were collected or assessed for this study.
Arm/Group | Population Health Management | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/37/NCT03077737/Prot_SAP_000.pdf